CLINICAL TRIAL: NCT05406518
Title: Proposal to Improve the Program of Attention to the Families of the Community Rehabilitation Service "Dr. Pi i Molist": Implementation and Evaluation Based on a Needs Analysis
Brief Title: Proposal to Improve the Program of Attention to the Families. Implementation and Evaluation Based on a Needs Analysis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Collaborators: University Ramon Llull (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIBSP-PAF-2021-70
Record Dates: First submitted 2022-06-02; First posted 2022-06-06 (Actual); Last update posted 2022-06-06 (Actual); Status verified 2022-06

CONDITIONS: Severe Mental Disorder
Keywords: family; psychosocial; rehabilitation
MeSH Terms: conditions — Mental Disorders | interventions — Psychosocial Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Arm of intervention
  Interventions: Other: Psychosocial intervention

INTERVENTIONS:
Other: Psychosocial intervention — Psychosocial intervention based on the model of family therapy.

SUMMARY:
Applied research carried out in the context of the Community Rehabilitation Service "Dr. Pi i Molist". The objective is to improve the psychosocial intervention carried out with the families of the patients treated (Severe Mental Disorder). It is proposed to carry out a qualitative needs analysis with relatives, patients and professionals, with the intention of detecting possibilities for improvement. With the results obtained, together with the bibliographic recommendations, a new intervention proposal is made and the new results obtained are evaluated. The hypothesis is that a form of intervention more adjusted to the real needs of the population and more effective for the engagement of families and the improvement of the quality of life of patients and their families can be found.

DETAILED DESCRIPTION:
1. THEORETICAL FRAMEWORK. PROBLEM STATEMENT

   1.1 Conceptualization

   Severe Mental Disorder (TMS) is defined from the confluence of three criteria: a clinical diagnosis of mental health considered one of the most serious, a high affectation or duration and a high presence of disability at the functional level (National Institute of Mental Health [NIMH], 1987; Servei Català de la Salut, 2003a). Its prevalence is between 3-5% of the general population (Gaebel et al., 2016; Ministry of Health, 2017; NIMH, 2019).

   One of the main treatments for people with TMS is Psychosocial Rehabilitation (RPS), as reflected in most Clinical Practice Guidelines (American Psychiatric Association [APA], 2020; Ministry of Health and Consumer Affairs, 2009; National Institute for Health and Care Excellence [NICE], 2014) and in the recommendations of the administration (Generalitat de Catalunya, 2017; (World Health Organization [WHO], 2013).

   The RPS is defined, rather than as a set of techniques, as a philosophy of care (Leal & Castilla, 2002; Vazquez et al., 2000) whether to conform rigidly to any model or strategy of intervention (Gisbert, C; Arias & Campus, 2002). Currently the predominant model works on the idea of Recovery (Pérez, 2012) which highlights the importance of highlighting psychosocial aspects over purely clinical ones (Anthony, 1993) and the active role of users in their improvement process (Deegan. 1988).

   Community Rehabilitation Services (CRS) are health resources, sectorized and dependent on the Mental Health and Addictions Network, oriented to the care of people with TMS (Servei Català de la Salut, 2003b). CRS are considered the backbone and coordinator of Psychosocial Rehabilitation (PRS) treatments (Generalitat de Catalunya, 2007). According to the Servei Català de la Salut (2003b) family intervention is one of the basic intervention programs of an SRC.

   The SRC Dr. Pi i Molist, the first to be inaugurated in Catalonia (Grup de Treball de Serveis de Rehabilitació Comunitària, 2006), is located within the Dr. Pi i Molist Community Resources Unit, depending on the Psychiatry Service of the Hospital de la Santa Creu i Sant Pau. It has 104 public assistance places for people with TMS and is integrated into the Mental Health Circuit of Nou Barris (Barcelona).

   1.2 Theoretical foundation The beginning of the study of the family of people with a TMS in the early twentieth century can be placed within the school of psychoanalysis, but with a causal interpretation and without proposals for intervention beyond the individual with the affected patient (Fallon et al., 1996). In the mid-50s of the twentieth century, Systemic Family Therapy appeared, assuming a paradigm shift that questions the linear causality of cause and effect (Nardone & Watzlawick, 1995). According to this vision, the family is defined as a system (Botella and Vilaregut, 2010) and the patient as part of a complex system, its symptoms being able to be explained according to the dynamics of the system (Feixas et al., 2016). Although the systemic model has remained the most widespread conceptual framework in terms of family intervention (Feixas et al., 2016) and there is evidence that it remains so with respect to people with TMS (Gaebel et al., 2016; Pharoah et al., 2010; Petersen et al., 2005, cited in Sempere, 2015; Rangel, 2019) was losing popularity with respect to intervention in this population and replaced in the 70s by simpler models (Linares, 2019).

   Brown et al. (1972) managed to define the components in terms of family attitudes more linked to relapses and, from this, Leff and Vaughn (1976) created the model of Expressed Emotion (EE). This model is purely clinical, without a complex theoretical basis, and perhaps that is why it could be generalized more easily (Touriño et al., 2004). Some criticism he received was, for example, not to pick up the discomfort and overload of families, which proved to be high and generate disability (Magliano et al., 1998; Rangel, 2019; Schulze & Rössler, 2005).

   From the end of the twentieth century and the beginning of the twenty-first century, generally recovering a broader theoretical base, multifamily groups for people with TMS became popular (Sempere, 2015). There are models that are especially relevant such as the one proposed by Fallon (Fallon et al., 1995) or the Open Dialegue (Seikkula, 1994; Seikkula et al., 1990), but the one that acquires greater popularity the proposal of McFarlane, since it obtains very high efficacy data (McFarlane, 2016) with ease to be replicated (Sempere & Fuenzalida, 2017). Its proposal is of groups where users and relatives participate and with a special attention to the engagement and linkage (McFarlane, 2002).

   The therapeutic joining of families (Minuchin, 1974), also sometimes called family alliance (Escudero, 2009) is assumed by many authors as a frequent difficulty regarding treatment, being necessary to address it specifically (Beck et al., 2006; Escudero, 2009; Karin et al., 2010; Linares, 2012; Friedlander et al., 2009; Friedlander et al., 2006). In the context of RPS, the lack of engagement or linkage is also considered as a common difficulty that requires specific interventions (Gisbert, C; Arias & Campus, 2002; González & Rodríguez, 2002; IMSERSO, 2007; Perez, 2012; Vargas & Touriño, 2010), even specific for family members (Gisbert, 2003; Touriño et al., 2004).

   1.3 Justification Family intervention in people with TMS, in its different modalities, has been shown to be consistently effective (Pharoah et al., 2010; Pilling et al., 2002; Pitschel-Walz et al., 2001) and is a recommendation of the main clinical practice guidelines (Navarro, 2011).

   According to the Servei Català de la Salut (2003b), family intervention is one of the basic programs of an SRC. The same document also defines the Family Intervention Program (PAF), although it does not specifically specify the form of intervention, offering flexibility to each SRC, but single-family interventions, multifamily interventions, psychoeducational groups, problem-solving groups or standardized family intervention programs are mentioned as possible recommended activities (Generalitat de Catalunya, 2007). Authors point out that the lack of family intervention may be one of the main reasons why people do not improve in their RPS treatments (Leal & Castilla, 2002; Navarro, 2011).

   The SRC Dr. Pi i Molist has an active PAF that defines single-family and multi-family interventions. The engagement of single-family interventions seems adequate (in 98% of family members some intervention was made during 2019), but not so in group interventions (average attendance in recent years of 6 relatives on a call of 70). Different models (psychoeducational models based on EE, monographs on RPS, open groups, self-help format, etc.) and strategies (recently incorporated relatives, longer, at different times, durations and frequencies, etc.) have been tested without detected improvement. Multifamily groups with the presence of users have never been carried out.

   Group intervention has advantages over single-family intervention. In addition to the most obvious, cost-effectiveness, for several authors has advantages such as improving socialization (Barbagelata, 2018), functioning and structuring (Fontes & Gabriela, 2014) or self-esteem, comparing, accepting reality, containing anxiety and inducing hope (Herández & Nieto, 2016) and, above all, favoring emotional expression with the help of others, so that it can be processed and managed (Sempere & Fuenzalida, 2017).
2. RESEARCH QUESTIONS. HYPOTHESIS. OBJECTIVES

   2.1 Research Questions What needs are currently not met and proposals for improvement do the participants of the SrPH Dr. Pi i Molist Family Care Program have? Will the new proposal arising from the expressed needs and proposals improve the engagement of families and help them and users to improve their quality of life?

   2.2 Hypothesis The needs of families not covered will be detected in the current PAF program of the SRC Dr. Pi i Molist.

   The new PAF programme will respond to the needs of the families served. The new PAF program will improve the therapeutic engagement of families. The new PAF program will improve the quality of life of users and families.

   2.3 Objectives Identify the needs and proposals for improvement by users, family members and professionals of the SRC Dr. Pi i Molist regarding the Family Care Program (PAF program).

   Design, implement and evaluate a new PAF program Assess whether the new proposal increases the therapeutic engagement Evaluate whether the new PAF program improves the quality of life of users and family members
3. METHOD

   3.1 Study design This study is presented as an applied research project, starting from a phenomenological and interpretative paradigm. It presents two parts, one of analysis of the needs of a specific population from which an adapted intervention program will be developed, and another of evaluation of the results of the intervention and its influence on the improvement of the quality of life. To this end, a mixed methodology will be used, qualitative for the analysis of needs, and quantitative for the evaluation of the intervention.

   In the preparation of the new intervention proposal, a series of actions are proposed, following the scheme recommended by Anguera et al. (2008) regarding the development of programs.

   According to this proposal, the SRC Dr. Pi i Molist is currently towards the end of the process, having a program, the PAF, already developed and in the intervention phase. However, the needs do not seem to be being met according to the opinion of the SRC management and the professionals involved, but it can also be the message that the families themselves transmit with the lack of engagement and assistance to the groups.

   Based on the design described, a series of 3 phases are proposed with actions to be carried out to carry out the elaboration of the new PAF of the SRC Dr. Pi i Molist. Previously, coordination has been carried out with the center where the project will be carried out, the SRC Dr. Pi i Molist, ensuring its acceptance by the management, adjusting the demand and favoring the collaboration of the agents involved.

   The first phase will focus on analysis for the detection of needs. It will be made from the src database Dr. Pi i Molist, from a list of possible participants for the focus groups. To make the call, the telephone call will be used, explaining the project and requesting your initial interest to participate. If the answer is yes, they will be summoned individually by the researcher to explain the study in more detail, ensuring understanding of it, checking if the inclusion / exclusion criteria are met and requesting the acceptance and signature of the informed consent. After that, they will be asked to fill out the sociodemographic questionnaire where an alphanumeric code corresponding to each participant will be assigned.

   When the groups are formed, they will be programmed in the same space as the Dr. Pi i Molist center and will be led by a researcher who will try to follow the script with a flexible format, promoting debate, interaction between members and the emergence of new information. The duration of the group will be approximately one and a half hours. Focus groups will be recorded in audio and then anonymized, encoded and transcribed into text.

   Due to the current context of the COVID-19 pandemic, it is possible that focus groups will have to be done online. For this, the Google Meet computer suite would be used.

   The second phase corresponds to the development of the new PAF. The information obtained in the previous step will be analyzed and contrasted with the scientific literature. A new intervention program will be developed taking into account criteria of acceptability for stakeholders, adequacy, quality, coherence, efficiency, utility, ethics and viability (Anguera et al., 2008), but also considering as a priority the adjustment to the specific population and the needs and proposals that the participants have made.

   In this phase, the sections recommended by Fernández-Ballesteros (1992) for the elaboration of programs will be followed, assessing whether there are elements of the previous program that can fit into the new proposal, which should be reviewed and which incorporated again.

   Although some of the proposed stages are already defined in this plan, they will also be reviewed, assessing their suitability for the new program. The new program will be presented to the management and workers of the center, seeking their complicity and collaboration in it. In the design of the new PAF, the different actions and evaluation methods that will be applied in this phase will have been defined, using appropriate and rigorous tools, also ensuring that they are commonly used in the RPS environment. The design will include a further review of methodology, ethics and the development of a new informed consent to be used.

   Finally, in the third phase, the new intervention proposal will be implemented and its results will be evaluated. At this stage, the interventions foreseen in the new PAF and the selected evaluation methods will be applied. Subsequently, the data will be analyzed and the final document of results and conclusions will be elaborated, promoting its dissemination through its publication.

   3.2 Study population. Following the recommendations of Morgan (2019) for the focus groups, it will be ensured that they present internal homogeneity, that is, that the members of the groups have similarities between them in relation to the research topic, but at the same time there is greater heterogeneity between groups, so that they collect a greater number of perspectives. For the topic that interests us, the needs of family intervention in the SRC Dr. Pi i Molist it is evident that the voice of the families will be relevant and from them a focus group will be constituted, but so will be the opinion of the users served in the resource and of the care professionals who work with the users and / or families.

   Therefore, 3 focus groups will be carried out: family members, users and professionals. As a common factor we will find the size that, following the recommendations of Morgan (2019) will be from 6 to 12 people. In the evaluation phase of the new intervention proposal, it will only be carried out with family members and users.

   3.2 Expected sample size For the needs analysis, 3 groups (users, family members and professionals) are expected, with a range of 6 to 15 participants. Therefore, the average would be about 9 participants per group and 27 participants in total, and the maximum of 45 participants.

   For the evaluation of the new intervention proposal the sample size cannot yet be defined as it depends on the results of the previous phase.

   3.3 Methodology. Sources of information This is a qualitative (needs analysis phase) and quantitative (evaluation phase of the new intervention proposal) mixed design.

   3.4 Data management and analysis Regarding the part of analysis and detection of needs, the data collected in the focus groups recorded in audio will be transcribed and analyzed according to the thematic analysis procedure proposed by Braun and Clarke (2006), which offers an approach approach to data that is characterized by accessibility and flexibility at the theoretical level. The process begins with the search for patterns of meaning and issues of potential interest from the information collected, the ultimate goal being to identify the patterns (themes) that emerge from the data. To help in the analysis process, the computer tool of qualitative analysis Atlas.ti in its version 9 will be used.

   To clarify the procedure Braun and Clarke (2006) propose a guide of six phases of analysis. However, the same authors insist on not following a purely linear process in which one simply advances from one phase to another, but by following a more recursive process, where the movement is back and forth as needed.

   Regarding the evaluation phase of the new intervention proposal, the quantitative data of the different scales administered will be analyzed. The sociodemographic and linking information, only collected at the beginning of the intervention, will be analyzed in a descriptive way. For the quantitative results of the other scales, statistical contrasts will be made to verify the effect of the intervention. For all these analyses, the IBM SPSS version 23.0 statistical package will be used.

   The person responsible for the creation of the database, data entry and statistical analysis will be Javier Piris Alonso, psychologist of the SRC Dr. Pi i Molist (Community Resources Unit Dr. Pi i Molist, Psychiatry Service, Hospital de la Santa Creu i Sant Pau)

   3.5 Quality control The researcher will guarantee the accuracy and completeness of the data, as well as all the reports that are required. The data included in the Data Collection Notebook (CRD), which are derived from source documents, will be consistent with said documents or otherwise the discrepancies will be justified.

   The researcher will keep the documents of the study until at least 5 years after its completion.

   At the request of the monitor, auditor, CEIC or health authority, the researcher will have available all the files related to the study, allowing direct access to the data or source documents for the monitoring, the audit, the review by the CEIC, as well as the inspection of the test by the competent authorities.

   3.6 Limitations of design, source of information and methods of analysis The project has some limitations of research in the human sciences, as well as being an applied research project. First, all the data will come from a single intervention center, since it is intended to adapt the intervention to this specific situation, so it could present problems in terms of the generalization of the results. However, this limitation is also in itself a strength, since the process can be generalizable to other centers (CRS are frequent resources in the public mental health network) that with similar difficulties could replicate it.

   On the other hand, it is possible that, due to the characteristics of the population, there are possible participants who do not meet the inclusion criteria due to difficulties of cognition, communication or organic risks, which could limit representativeness. Also with regard to groups carried out with professionals, despite having taken into account and tried to reduce the possible negative repercussions of their opinions by excluding members of the management from the groups, they may self-limit their responses. It would be appropriate to propose in future research methodologies that can overcome these limitations.

   In this regard, also in terms of possible lines of future research, the replication of the program in other centers and in other territories, as well as with other populations, is proposed. It would also be a very interesting possibility to carry out a longitudinal study that allows assessing the effectiveness of the program over time.
4. ETHICAL ASPECTS:

   For this project, the principles of biomedical ethics of Beuchamp and Childress (2011) of non-maleficence, beneficence, autonomy, justice and confidentiality are contemplated, the Deontological Codes of Psychology, both of Catalonia and of Spain (Official College of Psychologists of Madrid, 2015; Col·legi Oficial de Psicologia de Catalunya, 2015) and the Declaration of Helsinki in its latest version (2017) Regarding the principles, starting with that of non-maleficence or avoidance of damage, it has been taken into account that the risk at the physical level is reduced, since no invasive procedure will be performed. However, an attempt will be made to reduce the discomfort in the form of fatigue that the collection of data may entail, avoiding the collection of irrelevant information. At the level of psychological discomfort, it will be avoided to unnecessarily address areas that may produce negative feelings and, since it is not always possible to control it, researchers will be attentive to detect the possible discomfort and be able to offer them to talk to their clinical referents. At the social level, the calls will be reduced in time and space, so the risk of isolation or loss of roles will be reduced. On a spiritual level it is difficult that there can be risk since it is not a topic related to the objectives of the study.

   Regarding the principle of charity, this project proposes, on the one hand, to give their own voice to the people involved in the programs, so that later interventions can be made adjusted to their needs and therefore more beneficial, and on the other hand these the scientific literature consulted guides us that interventions in relatives of people with TMS are beneficial both for families and for the users themselves.

   As for the principle of autonomy, all participants will be invited to collaborate voluntarily, freely and informedly. Particular emphasis will be placed on ensuring adequate understanding of the information on the study through a detailed explanation of the study orally and in writing and the use of clear and accessible informed consent. Sufficient time and space will be offered for you to ask questions and researchers will be proactive (confirmation questions) to ensure that no doubts have been left in the participants. In the case of people in a situation of legal guardianship, the consent of both the person and the guardian will be requested. All persons will have the possibility to revoke consent and not to continue with the investigation at any time.

   The principle of justice will be addressed by treating all participants equitably, especially those who may present the most difficulties. A possibly expected difficulty is in terms of comprehension and expression problems (either due to cognitive problems or language problems, in the case of migrants), so a clear, leisurely language will be offered, making clarifications if difficulties are detected, offering sufficient space and time and an adequate rhythm.

   Finally, confidentiality will be respected, as described in the informed consent (see appendix), through Organic Law 3/2018 on the protection of personal data and digital rights. All participants' data will be anonymized by means of an identification code, dispensing with their identification data regarding the collection and processing of their responses.

   They have also been taken into account both the deontological code of psychology of Catalonia (Col·legi Oficial de Psicologia de Catalunya, 2015), and the code of ethics of the psychologist of Spain (Official College of Psychologists of Madrid, 2015) that also collect some principles and a series of articles oriented exclusively to research.

   One of the principles is that of responsibility and, in this sense, the project will be carried out by specialist professionals trained and accredited to carry out both research and intervention. The study is led by a PhD in Psychology from the Faculty of Psychology, Education and Sports Sciences of Blanquerna (Ramon Llul University), has the approval of the management of the SRC Dr. Pi i Molist and will be evaluated before its start by the Ethics and Credentials Committee of the Hospital de la Santa Creu i Sant Pau.

   It also highlights the principle of integrity, by which in this research we will base relationships with participants on respect and honesty.

   Reference is made to the principle of legality, which is why this project complies with national and regional legality, taking special care regarding the treatment and protection of data, complying with the laws mentioned above.

   Regarding the investigations, particular reference is made in articles 45 to 49 in the Catalan version, and from 33 to 38 in the Spanish version, resulting in the content of the same very similar. We believe that at the ethical level these issues are resolved by compliance with the above principles and the attached informed consent. The rest of the articles refer to sections (studies with hidden objectives, animal experimentation or teaching) that do not apply in this project.

   Finally, we specify that it is not necessary to take out insurance, since the possibility of damages is practically nil. Nor does the payment or compensation to volunteers since it does not fit into the proposed methodology.

   Regarding the Declaration of Helsinki (2017), most of the proposed principles are also reflected in the previous points. It highlights, however, principle 23, by which there is a commitment to present and approve by a relevant Ethics Committee, prior to the start of the research. This protocol will be presented, pending advice, guidance and approval to the Clinical Research Ethics Committee of the Hospital de Sant Pau. Likewise, any subsequent modification of the protocol will be notified and subject to evaluation by this same committee.

   4.1 Ethical considerations, on information to the subjects and informed consent The study will be conducted in strict compliance with international ethical recommendations for medical research in humans. The researcher shall be responsible for ensuring that the study is carried out in accordance with the rules set out in the Declaration of Helsinki.

   Before starting the study, the Ethics Committee of the Hospital de la Santa Creu i Sant Pau must approve the study protocol, the information that will be given to the subject and the informed consent model that will be used.

   The CEIC will be informed of any subsequent amendments to the protocol and its opinion should be sought in the event that a re-evaluation of the ethical aspects of the study is necessary.

   It is the responsibility of the investigator to obtain the patient's informed consent. The patient will not be able to participate in any specific study procedure before obtaining their consent, or that of their legal guardian/family member when the patient is unable to give consent due to their clinical situation.

   Before including any subject in the study and before obtaining informed consent, the investigator or the person designated by the same, will explain to the potential participant subject or his legal guardian / family, the objectives, methods and potential risks of the study and any discomfort that it may cause. The explanation about the nature, scope and possible consequences of the study will be made in understandable language.

   The prospective participant or their legal guardian/family member will have sufficient time to ponder their decision to participate in the study, and have the opportunity to ask questions. After this explanation, and before entering the study, the consent must be properly recorded by the signature of the subject or his legal guardian / relative.

   The Model Patient Information Sheet and Consent Form of the first phase of the research are presented as an Annex. Since the explanatory information is identical for the three groups, the same model will be used for users, family members and professionals.

   As the specific format of the intervention phase will depend on the results of the first phase of needs analysis, a new information sheet and informed consent model will be prepared and sent to the Ethics Committee of the Hospital de la Santa Creu i Sant Pau before its application.

   4.2 Confidentiality of data Regarding the confidentiality of the data of the study, the provisions of Organic Law 3/2018, of December 5, on the Protection of Personal Data and Guarantee of Digital Rights and the General Regulation (EU) on Data Protection 2016/679 will be followed.
5. PLANS FOR THE DISSEMINATION OF RESULTS:

This project is part of the Doctoral studies of the Universitat Ramon Llull - Blanquerna. Therefore, the publication plans are framed within the doctoral program and, specifically, with respect to the thesis by compendium of publications, which requires the publication of at least three articles in journals that have an evaluation system by co-exembblants and indexed preferably in international scientific databases.

ELIGIBILITY:
1. Families: the call will be made with relatives of users currently linked to the SRC and with whom some type of contact has been previously established and who have been presented, both by the user and by themselves, as a reference relative. It is assumed that their similarities with the research topic (all will have a family member with TMS diagnosis who is carrying out an RPS process) will already generate sufficient homogeneity and it will not be necessary to perform a segmentation. Bear in mind that, as the age of some family members may be high or their health situation may be delicate, special care will be taken that their participation does not pose a clinical risk, something especially relevant in the current context of the COVID-19 pandemic. The following inclusion and exclusion criteria will be followed:

   Inclusion criteria
   * Be of legal age (18 years).
   * Have a family member cared for in the SRC with a minimum relationship of 3 months.
   * Have had previous contact with the SRC, having been presented as a family member of reference.
   * Understand, accept and voluntarily sign the informed consent.
   * Properly understand the reasons of the group and the project.

   Exclusion criteria
   * Present severe communication or cognitive problems that prevent the understanding of the questions or the possibility of participating in group communication.
   * It is assessed that, due to age or health situation, participation in the group may pose some clinical risk.
2. Users: those who are currently linked to the SRC and who have active family ties may participate. It is assumed that their similarities with the research topic (all will have relatives susceptible to being cared for by the SRC) will already generate sufficient homogeneity and it will not be necessary to carry out a segmentation. As one of the objectives of the SRC is to work on communication skills and some users may have deficits in these areas, it will be especially important to value having a minimum skill to be able to participate in the focus group properly. Also note that since the SRC Dr. Pi i Molist places in its "Program of reception and linkage", the time of incorporation to the center in 3 months, the participants of the focus group will be selected from that time of linkage. The following inclusion and exclusion criteria will be followed:

   Inclusion criteria
   * Be of legal age (18 years).
   * Minimum linkage in the SRC (more than 3 months).
   * Have previously presented a family member to the service as a reference relative.
   * Understand, accept and sign the informed consent.
   * Properly understand the reasons of the group and the project.

   Exclusion criteria
   * Present severe communication or cognitive problems that prevent the understanding of the questions or the possibility of participating in group communication.
   * It is assessed that, due to age or health situation, participation in the group may pose some clinical risk.
3. Professionals: will be those who perform direct assistance in the SRC Dr. Pi i Molist with users and / or relatives. Following the recommendations of Morgan (2019) for the realization of focus groups where members know each other and there may be hierarchical relationships, authority figures (director and coordinators) will not be included with whom, on the other hand, previous contacts have been made transmitting the institutional mandate that has given rise to this study, and they have been informed, their ideas and suggestions have been heard and integrated and this research plan has been approved. The greatest participation and representativeness of the participants will also be sought. Beyond this, the following inclusion and exclusion criteria are followed:

Inclusion criteria

* Perform tasks of assistance to users and / or relatives in the SRC.
* Minimum time in the SRC (more than 3 months).
* Understand, accept and sign the informed consent.
* Properly understand the reasons of the group and the project.

Exclusion criteria

- Management staff of the center.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-03-25 (Actual); Primary Completion 2022-04-26 (Actual); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Patients' family needs | 6 months
  Intervention needs in family members of users with severe mental disorders

CONTACTS AND LOCATIONS:
Locations (1):
- Fundació de Gestió Sanitària de l'Hospital de la Santa Creu i Sant Pau, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided